CLINICAL TRIAL: NCT06397261
Title: Artificial Intelligence Assisted Tracheal Video Intubation: an Observational Trial About Correctness of LarynGuide™
Brief Title: LarynGuide™ Assisted Tracheal Intubation
Acronym: LarynGuide
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: aiEndsoscopic (Unknown)
Responsible Party: Principal Investigator, Thomas Riva, Prof. Dr. med. Thomas Riva, Insel Gruppe AG, University Hospital Bern
Other Study IDs: LarynGuide
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-05

CONDITIONS: Intubation
Keywords: Artificial Intelligence; Tracheal video intubation; larynGuide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult patients undergoing elective surgery: adult patients undergoing elective surgery requiring tracheal intubation
  Interventions: Device: LarynGuide

INTERVENTIONS:
Device: LarynGuide — Artificial Intelligence assisted tracheal video intubation

SUMMARY:
This study aims to asses if the application of the larynGuide™, an assistive software running on a video-laryngoscope platform guiding laryngoscopy and intubation advise correctly and reliably on the position of the tracheal tube after an intubation attempt.

DETAILED DESCRIPTION:
Eligible patients will be prepared for intubation according to the local SOPs of the anesthesia departments with mandatory monitoring of SpO2, HR, NIBP, EtCO2.

For the anesthesia Patients will be pre-oxygenated before induction via face-mask with FiO2 = 1.0 and flow rates of 18L/min until etO2 reaches 90%. Induction of anesthesia and TI will be performed using a combination of sedative/hypnotic drugs, opioids and non-depolarizing muscle relaxant. The following medications will be mandatory as per protocol:

* Hypnotic agent (Propofol 1-4 mg/kg).
* Opioids (Fentanyl 1-3 mcg/kg, Remifentanyl 1-3 mcg/kg).
* Non-depolarizing muscle relaxant (Rocuronium 0.5-1 mg/kg). After induction of anesthesia and the administration of the muscle relaxant, bag-mask ventilation with FiO2 = 1.0 (flow rates of 18 Lmin-1) will be performed until apnea sets in. After induction all patients will be paralyzed to facilitate airway management. Neuromuscular blockade will be assessed by train-of-four monitoring. Thereafter oxygen administration, laryngoscopy and tracheal intubation are performed as usually.

Tracheal intubation performed with the aid of larynGuide™, an assistive software running on a video-laryngoscope platform guiding laryngoscopy and intubation (aiEndoscopic, Zürich, Switzerland). The larynGuide™ will be combined with the C-MAC video laryngoscope (Karl Storz, Tuttlingen, Germany) with a Macintosh nr 3 or 4 blade by a board-certified anesthesiologist. The board-certified anesthesiologist performing the intubation communicates to the research staff when he completed the intubation attempt. The anaesthesiologist in charge (board certified) checks to assess the correctness of the tube position by visual check and by attaching the patient to the ventilator and measuring the endtidal CO2 (Gold standard for detection of tube placement in anesthesia).

For the study the research staff will then - after the confirmation of the anaesthesiologist in charge of the tubes correct placement - look if the software displays a green light or the words "Bad intubation" on the monitor and document either outcome.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients ≥18 years
* ASA class I to III
* undergoing elective surgery in general anesthesia with tracheal intubation

Exclusion Criteria:

* Contraindication for intubation with C-MAC video laryngoscope (Karl Storz, Tuttlingen, Germany) with a Macintosh nr 3 or 4 blade
* Patients < 18 years
* No proper trained personnel for the device at the study site
* Expected impossible mask ventilation.
* High risk of aspiration (requiring rapid sequence induction intubation)
* Intracranial surgery
* Limited knowledge of German language or refusing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: german speaking adult patients classified ASA I, II or III undergoing surgery (except intracranial surgery) in general anaesthesia with tracheal intubation without contraindication for intubation with C-mac or indication for impossible mask ventilation and high aspiration risk with given informend consent.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Rate of correct assessment given by larynGuide™ | 5 minutes
  Correctness of the advice measured by accuracy of the LarynGuide™, a software for artificial intelligence assisted tracheal intubation (aiEndoscopic, Zürich, Switzerland) on tube position given at the end of an intubation attempt

SECONDARY OUTCOMES:
Overall success rate | 5 minutes
  Overall success rate under assistance with larynGuide™
first-attempt success rate | 10 minutes
  First-attempt oro-tracheal intubation success rate confirmed with waveform capnography in percentage
Number of attempts | 5 minutes
  number of attempts until correct intubation
Number of incidents of technical problems of larynGuide™ | 10 minutes
  Number of the occurrence of any technical problem of the larynGuide™, a software for artificial intelligence assisted tracheal intubation (aiEndoscopic, Zürich, Switzerland)
Percentage of glottic opening | 2 minutes
  Best percentage of glottic opening (POGO)
Rate of Cormack & Lehane Score from 1 to 4 | 2 minutes
  Cormack-Lehane classification is used to describe laryngeal view during direct laryngoscopy and can be divided into 4 grades of which 1 is the best (all of the glottis can be seen - so the best view) and 4 is the worste (not even the epiglottis is visible - worst view) the occurrence of which we will be counting.
Occurrence rate of airway management complications | 5 minutes
  Complications during and after airway management such oral/airway injury with bleeding, difficult bag-mask ventilation, emesis, aspiration of gastric contents, hypotension necessitating treatment, hypoxia causing bradycardia requiring chest compressions, pneumothorax and the administration of resuscitation drugs

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riva, Prof., Principal Investigator — Bern Univerisity Hospital
Locations (1):
- Inselspital, Bern, Canton of Bern, Switzerland